CLINICAL TRIAL: NCT02751411
Title: Multicenter, Prospective, Comparative, Randomized Controlled Clinical Trial to Evaluate the Performance and the Safety of Promelaxin® Micro-enemas Vs. Macrogol 4000 Per os in the Treatment of Functional Chronic Constipation in Children Aged Between 6 and 48 Months.
Brief Title: Effectiveness & Safety of Promelaxin® Microenemas Against Macrogol 4000 P.O. in Chronic Constipation in Children 6-48 Months
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Eclisse - Euromed Clinical Supply Services Srl (Unknown); Ceinge - Biotecnologie Avanzate s.c. a r.l. (Unknown); Latis S.r.l. (Industry); PhAST Consulting Srl (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABO-MELI-15
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Chronic Functional Constipation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: Randomized between two treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- micro-enema with Promelaxin (Experimental): 2,5 g, 5 g or 2X5 g (calculated considering patient age) have to be administered daily (in the evening) for one week, once every other day for the second week and as needed for the following 6 weeks
  Interventions: Device: micro-enema with Promelaxin
- Macrogol 4000 (Active Comparator): One/Two sachets of the study treatment has to be solubilized in 50mL of water and then administered daily. The administration should take place in the morning (the first sachet or in the event that only one sachet/day should be administered) and in the evening (second sachet).
  Interventions: Drug: Macrogol 4000

INTERVENTIONS:
Device: micro-enema with Promelaxin — The intervention has a lubricating, protective action on the anus and rectum and a balanced osmotic action which elicits the evacuation reflex.
  Other Names: Melilax
  Arms: micro-enema with Promelaxin
Drug: Macrogol 4000 — Stool softener
  Other Names: Paxabel
  Arms: Macrogol 4000

SUMMARY:
The study is aimed at the efficacy and safety evalutation of the study treatments through a 2-weeks study period and the subsequent follow-up-

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, controlled trial will be conducted on 120 infants-children with a diagnosis of chronic functional constipation according to the definition of Criteria of Rome III. The enrolled subjects will be randomized according to an electronically generated randomization list in 2 groups: one group will receive micro-enemas of Promelaxin® (Group A) while the second group will receive Macrogol 4000 per os (Group B) . Children will receive the dedicated treatment for two weeks and then undergo a follow-up period of a maximun of 6 weeks.

The hypothesis is that the protective micro-enema will help achieving regular evacuation by its local antinflammatory non-pharmacological action. This hypothesis is based on the finding that local anal inflammation can cause functional constipation due to discomfort and pain during evacuation or by influencing reflexes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic functional constipation according to Rome III criteria
* No stool softeners therapy administered during the 7 days prior to Baseline Visit
* Signature of informed consent from by both parents or legal representative
* Willingness to follow the study schedule

Exclusion Criteria:

* Suspicious or established diagnosis of organic constipation
* Delayed emission of meconium in the term newborn
* Presence of severe inflammatory bowel disease (such as ulcerative colitis, Crohn's disease), toxic megacolon
* Presence/Risk of gastroinstestinal perforation
* Presence/Suspiceous intestinal obstruction of symptomatic stenosis
* (Undeterminated) Abdominal pain
* Hypersensitivity to macrogol (polyethylene glycol) or to one or more product excipients
* Hereditary fructose intolerance
* Known hypersensitivity or allergy to any Promelaxin component
* Presence of any other medical condition that contraindicate the use of Promelaxin® or Macrogol 4000

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Improvement of constipation evaluated as a reduction of the typical symptoms of chronic functional constipation | day 14
  Treatment should be considered as successful if the child will show, at Visit 3, 3 or more defecations per week associated with an increase of 1 or more defecations versus baseline.

SECONDARY OUTCOMES:
score of the parents quality of life calculated on day 21 and 56 | day 21 and day 56
  parents quality of life questionnaire
score of the children quality of life calculated on day 21 and 56 | day 21 and day 56
  children quality of life questionnaire
Gastrointestinal symptoms in children on days 14, 21 and 56 | day 14, day 21 and day 56
  gastrointestinal symptoms recording through/following treatment
changes in the intestinal microbioma on day 21 and 56 | day 21 and day 56
  the intestinal microbioma will be analysed in laboratory to see whether a treatment influence can be measured
Evaluation of the normalization of intestinal activity measured by recording frequency of evacuations and stool consistency on day 14, 21 and 56 | day 14, day 21 and day 56
Product Safety | day 14, day 21 and day 56
  Adverse events reported by parents/legal representative of the subject
Change in stool consistency | day 14, day 21 and day 56
  Reduction of stool consistency with increase of 1 or more points on Bristol Stool Form Scale or Amsterdam scale

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Staiano, Prof., Principal Investigator — Universita Federico II - Pediatric Department
Locations (4):
- Italy (4):
  - ASL 1 Avezzano Sulmona L'Aquila - Ospedale San Salvatore - UO Clinica Pediatrica - Località Coppito, L’Aquila, AQ
  - Fondazione IRCCS Policlinico San Matteo di Pavia- Dipartimento Scienze Clinico-Chirurgiche, Diagnostiche e Pediatriche - Viale Golgi, 19, Pavia, PV
  - Dipartimento di Scienze Mediche Traslazionali - Pediatria - Università Federico II, Napoli
  - AOU Università degli Studi della Campania "Luigi Vanvitelli", Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strisciuglio C, Coppola V, Russo M, Tolone C, Marseglia GL, Verrotti A, Caimmi S, Caloisi C, D'Argenio V, Sacchetti L, Staiano A. Promelaxin Microenemas Are Non-inferior to Oral Polyethylene Glycol for the Treatment of Functional Constipation in Young Children: A Randomized Clinical Trial. Front Pediatr. 2021 Oct 29;9:753938. doi: 10.3389/fped.2021.753938. eCollection 2021. PMID 34778144